CLINICAL TRIAL: NCT05765435
Title: Effects of an Electrical Stimulation Program on Strength, Functional Capacity, Pain, and Gait in Individuals With Knee Osteoarthritis
Brief Title: A 12-Week Home-Based Electrical Stimulation Program for Strength in Adults With Knee Osteoarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient rate of accrual.
Sponsor: Cionic, Inc. (Industry)
Responsible Party: Principal Investigator, Rebecca Webster, Director of Clinical Operations and Research, Cionic, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIONIC-05-001
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Control (Other): Device: Cionic Neural Sleeve NS-100. Participants will wear the device during the 12-week exercise and walking program. There will be no stimulation.
  Interventions: Other: 12-week exercise and walking program
- NMES (Experimental): Device: Cionic Neural Sleeve NS-100. Participants will wear the device during the 12-week exercise and walking program and receive stimulation assistance during the exercise sessions.
  Interventions: Other: 12-week exercise and walking program; Device: NMES
- NMES and FES (Experimental): Device: Cionic Neural Sleeve NS-100. Participants will wear the device during the 12-week exercise and walking program and receive stimulation assistance during the exercise and walking sessions.
  Interventions: Other: 12-week exercise and walking program; Device: NMES; Device: FES

INTERVENTIONS:
Other: 12-week exercise and walking program — The exercise program requires isometric quadriceps contractions in a supine position with a rolled-up towel placed behind the knee. The exercise program will be performed by participants 5 days per week for 12 weeks. The walking program will be performed 3 days per week for 12 weeks. Participants will walk for 10 minutes and then gradually increase walking time to 30 minutes by the end of the study. Participants will wear the device during the exercise and walking program, which may range from 1 minute to 35 minutes per day.
Device: NMES — Sleeve applies neuromuscular stimulation during exercises to help contract appropriate muscles at appropriate times.
  Other Names: External functional neuromuscular stimulator
  Arms: NMES; NMES and FES
Device: FES — Sleeve applies functional electrical stimulation as patients walk to help contract appropriate muscles at appropriate times.
  Other Names: External functional neuromuscular stimulator
  Arms: NMES and FES

SUMMARY:
The purpose of this research is to investigate if a 12-week program of stimulation assisted activities can combat disuse atrophy for individuals diagnosed with knee osteoarthritis (KOA). This study will use a home-based medical device to administer electrical stimulation and measure its effect on outcomes that include quadriceps strength, perceived functional capacity, pain, and walking performance. It was hypothesized that stimulation assisted activities will show larger muscle mass and strength improvements; improved gait kinematics, pain and perceived function; and a high compliance to the assigned program compared to no stimulation.

DETAILED DESCRIPTION:
The study aims to evaluate the Cionic Neural Sleeve for subjects diagnosed with KOA. All participants will be assigned a Cionic Neural Sleeve to wear on the most impacted leg and be prescribed a home-based exercise and walking program. Participants will be randomly assigned into three groups: (a) control; (b) neuromuscular electrical stimulation (NMES); (c) NMES and functional electrical stimulation (FES). The control group will not receive stimulation for the exercise and walking program, whereas participants in the NMES group will receive stimulation during exercises, and participants in the NMES and FES group will receive stimulation during exercises and walking. The primary outcome measures include quadriceps strength and perceived pain. Exploratory outcome measures include adherence to the program, thigh muscle volume, functional ability of the lower limb, walking performance, perceived functional capacity, and perceived quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Persons with knee osteoarthritis between the ages of 22 and 75
2. Ability to walk a duration of 30 minutes per walking session (with or without an assistive device), for three days per week
3. Able to tolerate the device for up to 1 hour per lab session
4. No recent change in medication or exacerbation of symptoms over the last 60 days
5. Radiographic KOA Kellgren and Lawrence grade 2 or 3 or physician diagnosed mild or moderate KOA if radiographic imaging is not available
6. No hyaluronic acid or cortisone injection into knees in previous 12 months

Exclusion Criteria:

1. Lower motor neuron disease or injury (e.g. peripheral neuropathy) that may impair response to stimulation
2. Absent sensation in the impacted or more impacted leg
3. Inadequate response to stimulation, as defined as inability to achieve muscle contraction or tolerate stimulation
4. Inability to ambulate with the sleeve in place of an ankle foot orthosis (AFO)/knee ankle foot orthosis (KAFO) if utilized
5. Use of FES devices in the past year
6. Demand-type cardiac pacemaker or defibrillator
7. Malignant tumor in the impacted or more impacted leg
8. Existing thrombosis in the impacted or more impacted leg
9. Fracture or dislocation in the impacted or more impacted leg that could be adversely affected by motion from stimulation
10. History of knee replacement surgery
11. History of other types of arthritis
12. History of neurological disease
13. History of seizures or diagnosed with epilepsy/seizures
14. Current pregnancy

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cionic, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | NMES | NMES and FES
Started | 2 | 2 | 2
Completed | 2 | 1 | 1
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | NMES | NMES and FES | Total
Number analyzed (Participants) | 2 | 1 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 1 | 4
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 2 | 1 | 1 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Severity of Knee Osteoarthritis [Count of Participants; unit: Participants] — Population: Two subgroups, mild and moderate ...
  Participants
    Mild Severity of the Instrumented Leg | 2 | 0 | 0 | 2
    Moderate Severity of the Instrumented Leg | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Maximal Voluntary Isometric Contraction of the Quadriceps From Baseline
Description: Strength assessment of the quadriceps muscles using a handheld dynamometer, measured in Newtons. Subjects performed 3 repetitions of maximal effort, separated by two minutes of rest between each. The average of the 3 repetitions was recorded as the subjects' 1 repetition maximum. A positive change indicates increased quadriceps strength.
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Full Range); unit: Newtons
Arm/Group | Control | NMES | NMES and FES
Number analyzed (Participants) | 2 | 1 | 1
Newtons
  Change in Quadriceps Strength From Baseline to Week 6 | 76.62 [69.10 to 84.13] | 70.23 [70.23 to 70.23] | 148.47 [148.47 to 148.47]
  Change in Quadriceps Strength From Baseline to Week 12 | 76.38 [22.23 to 130.53] | 79.90 [79.90 to 79.90] | 198.90 [198.90 to 198.90]

2. Primary Outcome: Change in Perceived Pain Scores From Baseline
Description: Western Ontario/McMaster Universities Osteoarthritis Index (WOMAC) pain questionnaire to measure perceived pain, measured by score. Scores on the WOMAC pain subscale range from 0 to 20, with high scores indicative of worse pain. A positive change indicates improvement.
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Control | NMES | NMES and FES
Number analyzed (Participants) | 2 | 1 | 1
score on a scale
  Change in Pain From Baseline to Week 6 | 0.5 [0 to 1] | -1 [-1 to -1] | 1 [1 to 1]
  Change in Pain From Baseline to Week 12 | -2 [-5 to 1] | 0 [0 to 0] | 5 [5 to 5]

3. Other Pre Specified Outcome: Change in Perceived Functional Capacity
Description: WOMAC physical function (WOMAC-PF) questionnaire to measure perceived functional capacity, measured by score. Scores on the WOMAC-PF subscale range from 0 to 68, with high scores indicative of worse functional limitations.
Time Frame: Baseline, 6 weeks, 12 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Walking Performance
Description: Measured by gait speed via the 10-meter walk test (meters per second) and walking endurance via the 6-minute walk test (meters).
Time Frame: Baseline, 6 weeks, 12 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Adherence to the Program
Description: Measured by the usage log of the device or exercise diary/calendar, measured in minutes.
Time Frame: Daily
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Thigh Muscle Volume
Description: Measured by thigh circumference using a tape measure and prediction model to estimate muscle volume, measured in cubic centimeters.
Time Frame: Baseline, 6 weeks, 12 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Functional Ability of the Lower Limb
Description: Measured by the Five Times Sit to Stand Test, measured in seconds.
Time Frame: Baseline, 6 weeks, 12 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Perceived Quality of Life
Description: Short Form 36 questionnaire to measure quality of life, measured by score. Score ranges from 0 to 100, with 0 representing extreme interference, and 100 representing no interference in quality of life.
Time Frame: Baseline, 6 weeks, 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Control | NMES | NMES and FES
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT05765435/Prot_SAP_001.pdf